CLINICAL TRIAL: NCT02765139
Title: Preventing Intimate-partner Violence: Impact Evaluation of Engaging Men Through Accountable Practice in Eastern DRC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: World Bank (Other)
Collaborators: International Rescue Committee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P149394
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2018-05-21 (Actual); Status verified 2018-05

CONDITIONS: Intimate Partner Violence; Domestic Violence; Family Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMAP Treatment (Experimental): Engaging Men through Accountable Practice: 30 communities are matched into 15 pairs on a set of socio-demographic characteristic and within each pair, 15 treatment sites are randomly selected. Within each treatment community, all adult men (20+ years old) are eligible to participate in the EMAP intervention. A random draw of 50 participants determines who will participate in EMAP in case more than 50 eligible men express interest.
  Interventions: Behavioral: Engaging Men through Accountable Practice
- Control (Other): In the 15 control sites, the male participants will receive an alternative intervention focused on a non-gender topic of 16 weekly sessions for men only.
  Interventions: Other: Alternative intervention

INTERVENTIONS:
Behavioral: Engaging Men through Accountable Practice — Engaging Men through Accountable Practice aims to engage men as agents of change through structured, weekly discussions with committed groups of men. It aims to address entrenched views of gender roles and identify positive models of masculinity. The approach follows a structured series of discussions designed to explore existing understandings of masculinity and create more positive models of what it means to be a 'good' man, promoting self-reflection and pushing men to analyze and change their own power and privilege. This methodology begins with a series of discussions with women to inform men's dialogue groups, and includes continuous feedback loops with women throughout the process so that the work with men is grounded in, and accountable to, women's views and objectives.
  Arms: EMAP Treatment
Other: Alternative intervention — Control communities will receive an alternative intervention focused on a non-gender topic of 16 weekly sessions for men only.
  Arms: Control

SUMMARY:
The objective of the study is to evaluate the impact of Engaging Men in Accountable Practice (EMAP) on the prevention of violence against women and girls in North and South Kivu (DRC). The study is conducted jointly by the World Bank's Africa Gender Innovation Lab and the International Rescue Committee (IRC). EMAP is a program developed and implemented by the IRC to engage men to reflect on how to reduce and prevent intimate partner violence through 16 weekly group discussion sessions. The study is a cluster randomized control trial in which two groups of 25 self-selected men in 15 communities receive the EMAP intervention while in 15 other communities, 50 self-selected men receive an alternative intervention. Key outcomes examined include: (i) Experience of past year physical, sexual and psychological violence reported by women whose partners are EMAP participants; (ii) Participant's gender attitudes and behaviors, conflict and hostility management skills; (iii) Power sharing and communication within the couple.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 or older but preferably at least 25;
* Resident of their village, having lived in the community for a minimum of six months with plans to continue living there for at least the coming six months;
* Ability to participate actively in group work and reflection activities;
* Commitment to attend meetings, sessions and other activities regularly without incentives;
* Commitment to non-violence toward women and girls for the duration of the EMAP intervention;

Exclusion Criteria:

* Involved in the IRC-led adolescent girl intervention (COMPASS).

Min Age: 20 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1387 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in baseline prevalence of intimate-partner violence | Baseline, 12 months follow-up
  Change in the % of women who self-report experience of violence by their male partner. The women interviewed are the partners of the male study participants.

SECONDARY OUTCOMES:
Change in acceptability of intimate partner violence | Baseline, 12 months follow-up
  Change in the % of women (partners of participants) and men (participants) who report that violence is acceptable in at least one of the situations listed in the survey.
Change in intention to commit violence | Baseline, 12 months follow-up
  Change in the % of male participants who report that they are likely to become violent in a list of situations. Scale used: Proximal Antecedents to Violent Episodes.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Vaillant, PhD, Principal Investigator — World Bank
Locations (2):
- Democratic Republic of the Congo (2):
  - International Rescue Committee, Bukavu
  - International Rescue Committee, Goma

IPD SHARING:
Plan to Share IPD: Yes
The World Bank has an open data policy, and the de-identified, anonymized data will be published online after the study is completed.

REFERENCES:
- [Derived] Gurbuz Cuneo A, Vaillant J, Koussoube E, Pierotti RS, Falb K, Kabeya R. Prevention, Cessation, or harm reduction: Heterogeneous effects of an intimate partner violence prevention program in eastern Democratic Republic of the Congo. PLoS One. 2023 Mar 8;18(3):e0282339. doi: 10.1371/journal.pone.0282339. eCollection 2023. PMID 36888613
- [Derived] Vaillant J, Koussoube E, Roth D, Pierotti R, Hossain M, Falb KL. Engaging men to transform inequitable gender attitudes and prevent intimate partner violence: a cluster randomised controlled trial in North and South Kivu, Democratic Republic of Congo. BMJ Glob Health. 2020 May;5(5):e002223. doi: 10.1136/bmjgh-2019-002223. PMID 32467354